CLINICAL TRIAL: NCT06515054
Title: Effectiveness and Mechanisms of Isometric Resistance Exercise to Reduce Blood Pressure in a Chinese Population: a Pilot Randomized-controlled Trial
Brief Title: Isometric Exercise for Hypertension
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Lee Kam Pui, clinical associate professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRE001
Record Dates: First submitted 2024-07-15; First posted 2024-07-23 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-11

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension | interventions — Muscle Stretching Exercises

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- isometric exercise (Experimental): wall squat exercise. Each exercise session will contain 4 sets of 2-minute wall squat isometric holds with 2 minutes of rest between each set (approximately 14 minutes per session in total), and a total of 3 sessions will be arranged every week (with ideally 48 h between exercises)
  Interventions: Behavioral: wall squat
- passive stretching (Active Comparator): A frequency-matched (3x/week) and time-matched (~14 minutes each session) passive static stretching exercise will be used
  Interventions: Behavioral: passive stretching

INTERVENTIONS:
Behavioral: wall squat — self-learnt wall squat exercise to be conducted for totally 24 weeks
  Arms: isometric exercise
Behavioral: passive stretching — time-matched passive stretching exercise to be conducted for totally 24 weeks
  Arms: passive stretching

SUMMARY:
Background: Isometric resistance exercises (IREs) have great potential to improve blood pressure (BP) control.

Methods: This is a pilot randomized controlled trial that will involve 50 patients with hypertension (HT) who do not meet the current physical activity guidelines defined by the World Health Organization. Participants will be randomly assigned in a 1:1 ratio using stratified and blocked randomization to either the IRE (wall squat) group or stretching exercise (active control) group. A well-structured, widely accepted, and validated 24-week wall squat program (2 minutes per exercise, 2 minutes of rest between sets, and 3 sessions per week) will be implemented, as it has been commonly used in previous research. All patients will be followed up for 24 weeks. Control group will receive exact same treatment except that IRE is replaced by frequency-matched and time-matched stretching exercise. The primary outcome measure will be rate of recruitment. Secondary outcomes will include BP parameters from 24-hour ambulatory BP monitoring

ELIGIBILITY:
Inclusion Criteria:

* a suboptimal daytime SBP of >135-160 mmHg on a 24-h ABPM
* reported no regular physical activity or less than that recommended for adults by the World Health Organization (e.g. <150 minutes of moderate-intensity aerobic exercise per week);
* on stable doses of anti-HT medication(s) for ≥4 weeks if the patient is receiving drug treatments
* agree for no drug changes during the intervention period (24 weeks);

Exclusion Criteria:

* cannot provide informed consent
* unwillingness to repeat ABPM
* relative contraindications to ABPM (i.e. diagnosed atrial fibrillation, nighttime workers, occupational drivers, or patients with bleeding tendencies)
* severe osteoarthritis pending knee replacement surgery
* known secondary HT
* use of ≥3 anti-HT medications at maximum doses or ≥4 anti-HT medications
* SBP or DBP are >160 mmHg or >100 mmHg, respectively, on ABPM
* pregnancy/breastfeeding
* active malignancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2024-07-20 (Actual); Primary Completion 2025-09-30 (Actual); Study Completion 2025-11-30 (Actual)

PRIMARY OUTCOMES:
rate of recruitment | through study completion, an average of 1 year
  number of people recruited per month

SECONDARY OUTCOMES:
Blood pressure parameters | 24-week after recruitment
  24-hour, daytime and nighttime blood pressure from 24-hour ambulatory systolic and diastolic blood pressure measurement
Carotid-femoral pulse wave velocity | 24-week after recruitment
  analysed by applanation tonometry using SphygmoCor (AtCor Medical Pty Ltd) with the accompanying SphygmoCor Software Suite (SphygmoCor System)
flow-mediated velocity (FMD) | 24-week after recruitment
  FMD will be performed using a high-resolution linear artery transducer couple with a software (FMD suite, Quipu, Italy) that automatically detect and measure the brachial artery diameter and will be performed according to international guidelines

CONTACTS AND LOCATIONS:
Locations (1):
- School of public health and primary care, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Yes